CLINICAL TRIAL: NCT05728112
Title: Effectiveness Verification of Using Hydrogen Inhalation to Improve Fatigue, Pain and Quality of Life in Cancer Patients
Acronym: hydrogen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Collaborators: OTA HYDROGEN SOLUTIONS LTD. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KMUHIRB-F(I)-20210097
Record Dates: First submitted 2023-01-05; First posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2022-10

CONDITIONS: Head and Neck Cancer; Quality of Life; Pain; Sleep; Inhalation; Gas
Keywords: Head and Neck Cancer; Hydrogen; Cancer related symptom
MeSH Terms: conditions — Head and Neck Neoplasms; Pain; Respiratory Aspiration; Mucopolysaccharidosis IV

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrogen Inhalation (Experimental): The manufacturer installs the hydrogen inhalation machine at the subject's home and explains the relevant operation methods. The research executor will take care of it in the LINE group on the first day of installation, and after obtaining the pre-test baseline data (baseline data) through the google form, carry out each test. Continuous inhalation of hydrogen was carried out every day, and four post-test assessments were performed before inhalation and on the 1st, 3rd, 7th, and 14th days after inhalation.
  Interventions: Other: Hydrogen Inhalation
- Ordinary Air Inhalation (Placebo Comparator): This group used the same model to inhale, but the gas released was only ordinary air, as a placebo control.
  Interventions: Other: Ordinary Air Inhalation

INTERVENTIONS:
Other: Hydrogen Inhalation — The manufacturer will install a hydrogen inhalation machine (hydrogen inhalation or air inhalation) at the subject's home and explain the relevant operation methods. The research executor will pay attention to the LINE group on the first day of installation, and obtain the pre-test basic value data through the google form After (baseline data), continuous hydrogen inhalation was performed daily, and four post-test evaluations were performed before the inhalation and on the 1st, 3rd, 7th, and 14th days after the inhalation was started.
  Arms: Hydrogen Inhalation
Other: Ordinary Air Inhalation — The control group was inhaled with the same machine as the experimental group, but the gas was only ordinary air, which was used as a placebo control.
  Arms: Ordinary Air Inhalation

SUMMARY:
There are two recruitment methods for this study, which are mainly based on the Co-Principal Investigator Dr. Chih-Jen Huang recommendation of eligible subjects and poster recruitment methods.

When the subjects return to the outpatient clinic, those who meet the conditions for admission will be recommended by Dr. Chih-Jen Huang. If they agree to participate in the trial, they will sign the informed consent form, and instruct the subjects to use their mobile phones to scan the QR code of the relevant introduction of the trial first, and complete the test. The first questionnaire measurement before hydrogen inhalation; if the subjects are recruited by the poster, they can contact the host of Tongtong through the QR code on the poster or the contact number, and sign the consent form for the first time during the return visit. Questionnaire measurement.

DETAILED DESCRIPTION:
This study is a randomized controlled trial, and an experimental group and a waiting list group will be used to verify the interventional effect of hydrogen. For patients diagnosed with head and neck cancer who received radiation therapy or combined chemotherapy (CCRT) and met the inclusion criteria, the study was included after the study description and the consent of the trial were obtained. Investigators will be included, and the subjects will be numbered by the research executor (Co-Principal Investigator), and the number will be handed over to the project host, who will assign the subjects to the experimental group or the control group according to the random case allocation table generated in advance. The manufacturer will install a hydrogen inhalation machine (hydrogen inhalation or air inhalation) at the subject's home and explain the relevant operation methods. The research executor will pay attention to the LINE group on the first day of installation, and obtain the pre-test basic value data through the google form After (baseline data), continuous hydrogen inhalation was performed daily, and four post-test evaluations were performed before the inhalation and on the 1st, 3rd, 7th, and 14th days after the inhalation was started. The control group was inhaled with the same machine, but the gas was only ordinary air, which was used as a placebo control; after the experiment was over, if the moderator of the air inhalation group explained the plan, hydrogen inhalation would be given in the follow-up month for 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Adults over the age of 20
* Pathological diagnosed with head and neck cancer
* Received radiation therapy or combined chemotherapy
* Can use Mandarin or Taiwanese to communicate and have normal cognition

Exclusion Criteria:

* With chronic obstructive pulmonary disease
* Having contraindications to use of low flow oxygen
* Feeling uncomfortable using nasal cannula for inhalation

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline MDASI-Taiwan Form at 3rd days, 7th days, 14th days | Baseline, 3rd days, 7th days, 14th days
  Using MDASI-Taiwan Form: Divided into two parts, the severity of symptom distress and the degree of interference with life, a total of 19 questions, each question is scored from 0 to 10, 0 is no trouble, 10 is the most serious, and the average score after the evaluation is ≥4 Points indicate significant symptom distress.
Change from Baseline VSH sleep scale at 3rd days, 7th days, 14th days | Baseline, 3rd days, 7th days, 14th days
  Using Verran and Snyder-Halpern Sleep Scale(VSH sleep scale): It is divided into three subscales of sleep disturbance, effective sleep and compensatory sleep, with a total of 15 items. Using the visual analog measurement method using a 10 cm horizontal line, patients are asked to self-evaluate their feelings about sleep the night before and then evaluate their sleep patterns. There are 8 forward questions and 7 reverse questions in the questions. The minimum score for each forward question is 0 and the highest is 100 points. The opposite is true for the reverse questions. The overall sleep quality score is the sum of the total scores of the three subscales. In total, the total score ranges from 0 to 1500, with lower scores indicating poorer sleep quality.
Change from Baseline BFI-Taiwan Form at 3rd days, 7th days, 14th days | Baseline, 3rd days, 7th days, 14th days
  Using Brief Fatigue Inventory-Taiwanese (BFI-Taiwan Form): It is divided into five major items and nine sub-questions, including: whether there is unusual fatigue or fatigue in a week, the current level of fatigue, the general level of fatigue in the past 24 hours, the most fatigued level in the past 24 hours, and the impact of fatigue on life in the past 24 hours Level of influence, including: general activities, mood, ability to walk, normal work, relationships with others, enjoyment of life, etc. Each question is scored from 0 to 10, with 0 being no distress and 10 being the most serious, and the average of the scores after evaluation is ≥ 4, indicating significant symptom distress.
Change from Baseline European Quality of Life Scal-Five Dimensions Questionnaire (EQ-5D or EuroQOL) at 3rd days, 7th days, 14th days | Baseline, 3rd days, 7th days, 14th days
  Using EQ-5D: It is composed of two parts. In the first part, the subjects need to answer the health status of the day, including five questions: action, self-care, daily activities, pain/discomfort, and anxiety/depression. Each question has three options: "no problem", "some problem/moderate problem", "incapable of self-care/extreme problem", which can be weighted to get a single score. Five oriented questions can obtain 243 different health states, and through the group standard reference value established by time trade-off (TTO), a single EQ-5D score can be obtained after weighting (EQ-index ). The raw score on the EQ-5D was converted from -0.549 to 1, where 1 indicates "best state" quality of life, 0 indicates "death", and values below 0 indicate a state "worse than death".

CONTACTS AND LOCATIONS:
Overall Officials: YI-TSEN WU, Master, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan